CLINICAL TRIAL: NCT06958627
Title: The Impact of Intelligent Patient Management Model on Medication Adherence of Pyrotinib Compared to Traditional Patient Management Model: a Prospective, Multicenter, Randomized Controlled Clinical Study
Acronym: any
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Department of Medical Oncology, Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NCC4587
Record Dates: First submitted 2024-04-26; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: HER2 Positive Breast Cancer; Pyrotinib Treatment
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intelligent patient management model (Experimental)
  Interventions: Drug: pyrotinib
- traditional patient management model (Active Comparator)
  Interventions: Drug: pyrotinib

INTERVENTIONS:
Drug: pyrotinib — Intelligent patient management system on medication adherence of HER2 positive breast cancer patients receiving pyrotinib treatment.

SUMMARY:
This is a prospective, multicenter, randomized controlled clinical study to evaluate the effect of using intelligent patient management system on medication adherence of HER2 positive breast cancer patients receiving pyrotinib treatment. Pyrotinib is a small molecule tyrosine kinase inhibitor that can irreversibly inhibit HER1, HER2, and HER4.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years.
* Histologically confirmed HER2-positive breast cancer (IHC 3+ or IHC 2+ with ISH+).
* Patients expected to receive pyrotinib-containing regimens for neoadjuvant therapy or metastatic/unresectable breast cancer.

  ·≤1 prior line of anti-HER2 therapy during the recurrent/metastatic stage.
* Ability to operate a mobile phone and read independently.
* Deemed psychologically and physically suitable for participation by the investigator.

Exclusion Criteria:

* History of cognitive impairment.
* Severe visual or auditory impairments.
* Prior use of pyrotinib.
* Pregnancy, lactation, or intention to conceive.
* Ineffective cognitive-behavioral interventions within the past year.
* Participation in other clinical trials within 1 month prior to screening.
* Investigator judgment of unsuitability due to psychological or physical conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 964 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
medication adherence at 1-year | 1-year
  medication adherence at 1-year is assessed using the tablet counting method and Eight-Item Morisky Medication Adherence Scale Evaluation Method 1: Tablet Counting Method
  1. Definition/Formula:
     Adherence percentage = (Actual tablets taken / Total tablets prescribed) * 100% (Actual tablets taken = Total prescribed tablets - Remaining tablets - Lost tablets)
  2. Procedure:
  At the screening phase and Day 21 of each cycle, calculate the adherence percentage based on APP check-ins, and confirm the actual remaining tablets through follow-up.
  Evaluation Method 2: MMAS-8 Scale
  （1）Definition:
  The Morisky Medication Adherence Scale-8 (MMAS-8) is a validated 8-item questionnaire. The total score ranges from 0 to 8, with higher scores indicating better adherence:
  8: Good adherence 6-7: Moderate adherence <6: Poor adherence （2）Procedure: Administer the MMAS-8 scale at the screening phase and Day 21 of each cycle. The total score is calculated as the sum of scores from the 8 questions.

SECONDARY OUTCOMES:
The time to deterioration (TTD) | time from the date of randomization to the date of the first clinically significant deterioration through study completion, an average of 2 year
  TTD is defined as the time from randomization to confirmation of the first clinically significant deterioration (deterioration ≥ 10 points) in subsequent follow-up or death
Event-free survival (EFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  EFS (defined as the time from randomization to the first documentation of progressing disease while on study therapy, postoperative disease recurrence, or death from any cause)
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 4 years
  the time from randomisation to death from any cause
PRO | From date of randomization until the date of death from any cause, assessed up to 4 years
  EORTC QLQ-C30 and NCC-BC-A1.0 questionnaire：
  1. Outcome Measure 1 （1）Description: Scale Full Name: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
     Score Range:Global Health Status/QoL Scale: 0-100. Functional Scales (e.g., Physical, Role): 0-100. Symptom Scales (e.g., Fatigue): 0-100. （2）Interpretation: Higher scores on Global Health Status/QoL and Functional Scales indicate better outcomes.Higher scores on Symptom Scales indicate worse outcomes.
  2. Outcome Measure 2 （1）Description: Scale Full Name: National Cancer Center Breast Cancer-Specific Patient-Reported Outcome Scale Version 1.0 (NCC-BC-A1.0).
     Score Range:Total Score: 38-190 points (each item scored 1-5). （2）Interpretation:Higher total scores indicate poorer quality of life (for symptom-related items).Lower scores on positive function items (e.g., confidence, support) indicate worse outcomes.
  3. Time Frame: Baseline, every 2 cycles, and at end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jiani Wang, M.D., Principal Investigator — National Cancer Center Cancer Hospital
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD Description: Individual participant data will not be shared to protect patient privacy. The study involves sensitive clinical and behavioral data, and even de-identified datasets carry residual re-identification risks. Data access is restricted to the research team under ethical and legal obligations.
  Access Criteria: N/A IPD Sharing URL: N/A

REFERENCES:
- [Background] Koehler F, Koehler K, Prescher S, Kirwan BA, Wegscheider K, Vettorazzi E, Lezius S, Winkler S, Moeller V, Fiss G, Schleder J, Koehler M, Zugck C, Stork S, Butter C, Prondzinsky R, Spethmann S, Angermann C, Stangl V, Halle M, von Haehling S, Dreger H, Stangl K, Deckwart O, Anker SD. Mortality and morbidity 1 year after stopping a remote patient management intervention: extended follow-up results from the telemedical interventional management in patients with heart failure II (TIM-HF2) randomised trial. Lancet Digit Health. 2020 Jan;2(1):e16-e24. doi: 10.1016/S2589-7500(19)30195-5. Epub 2019 Dec 12. PMID 33328035